CLINICAL TRIAL: NCT03601052
Title: A Phase 2, Double-blind, Placebo-Controlled Study to Investigate the Efficacy, Safety and Tolerability of MRG-201 Following Intradermal Injection in Subjects With a History of Keloids
Brief Title: Efficacy, Safety, and Tolerability of Remlarsen (MRG-201) Following Intradermal Injection in Subjects With a History of Keloids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: miRagen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: MRG201-30-201
Record Dates: First submitted 2018-07-06; First posted 2018-07-26 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Keloid
Keywords: Keloid; MicroRNAs; Wound healing
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Intervention Model Description: Up to 6 cohorts of 12-16 subjects each may be enrolled to study various dose levels and dosing regimens.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The treatment administered to each of two wound sites will be randomized (left versus right), such that all subjects will receive both remlarsen and placebo in a double-blinded fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Remlarsen - Intradermal (Experimental): Six doses remlarsen (5.3 mg) over a period of 2 weeks at the site of one excisional skin wound and six doses Placebo over the same period at the site of a second excisional skin wound. Each subject will serve as their own simultaneous control.
  Interventions: Drug: Remlarsen
- Placebo - Intradermal (Placebo Comparator): Six doses remlarsen (5.3 mg) over a period of 2 weeks at the site of one excisional skin wound and six doses Placebo over the same period at the site of a second excisional skin wound. Each subject will serve as their own simultaneous control.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Remlarsen — Intradermal injection at site of one excisional wound
  Other Names: MRG-201
  Arms: Remlarsen - Intradermal
Drug: Placebo — Intradermal injection at site of second excisional wound
  Arms: Placebo - Intradermal

SUMMARY:
Remlarsen (MRG-201) is designed to mimic the activity of a molecule called miR-29 that decreases the expression of collagen and other proteins that are involved in scar formation. Remlarsen is being studied to determine if it can limit the formation of fibrous scar tissue in certain diseases. The objectives of this study are to investigate the safety and tolerability of remlarsen in subjects with a history of keloid scars, and to investigate the activity of remlarsen in prevention or reduction of keloid formation. Another objective is to study the pharmacokinetics of remlarsen (the movement of a drug into, through and out of the body). A group of 12-16 study volunteers will undergo two small skin biopsies in the upper back/shoulder region that will be closed with sutures. One biopsy site will be injected with up to 6 doses of remlarsen over a period of 2 weeks and the second site will be injected similarly with a placebo solution. Participants will be monitored for keloid formation at the two biopsy sites, for signs or symptoms of adverse effects on the body, and for the levels of remlarsen in the blood over time. A second 2-week cycle of treatment may be administered if there are signs that a keloid may be forming at one or both biopsy sites. Subjects will be followed for about 1 year following their final course of treatment to assess the long-term safety of remlarsen and the potential for later appearance of a keloid scar. Additional groups of subjects may be enrolled to test lower doses of remlarsen or an extended dosing schedule.

ELIGIBILITY:
Key Inclusion Criteria:

* Must provide written informed consent.
* Females must not be pregnant, or lactating, and have negative pregnancy tests.
* Study candidates should be likely to form keloids in the upper back/shoulder area after punch biopsy based on a history of a high frequency of keloid formation (≥ 10 keloids) or a history of large keloids (≥ 4 cm).
* Subjects should not anticipate requiring systemic corticosteroids during the study.
* Must have area in upper back/shoulder region free of keloids, acne, striae, or other skin pathologies or complications.
* Female subjects of childbearing potential or male subjects engaged in sexual relations with a female of childbearing potential must be willing to use a highly effective method of contraception throughout their study participation and for at least 6 months after the last dose of study drug.

Key Exclusion Criteria:

* Clinically significant abnormalities in medical history or physical exam that, in the opinion of the Investigator, would make the subject unsuitable for inclusion in the study.
* History of genetic disorders that predispose to keloids (e.g. Ehlers-Danlos syndrome, Ullrich congenital muscular dystrophy, etc.).
* History of renal or liver dysfunction or evidence of renal or liver dysfunction at screening.
* Evidence of clinically significant anemia, neutropenia, or thrombocytopenia at screening.
* History of bleeding diathesis or coagulopathy.
* Active or uncontrolled infection at screening or baseline.
* Recent history of alcoholism, drug abuse or illicit drugs (within the last year), and agreement to refrain from using illicit drugs throughout the study.
* Positive for bloodborne pathogen (HBV, HCV, HIV) at screening.
* Prior malignancies within the past 3 years (allowing squamous cell and basal cell carcinomas that have been successfully treated).
* Use of systemic steroids within 4 weeks of the Baseline visit or local use of steroids within 1 week of the Baseline visit.
* Use of an investigational small molecule drug within 30 days of the baseline visit or use of an investigational oligonucleotide or biologic drug within 90 days of the baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Escolar, MD, FAAN, Study Director — miRagen Therapeutics, Inc.
Locations (4):
- United States (4):
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - Northwestern University, Chicago, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - J & S Studies, College Station, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at four medical centers
Groups:
- Remlarsen-Treated Excisional Skin Wound and Placebo-Treated Excisional Skin Wound: Six doses remlarsen (5.3 mg) over a period of 2 weeks at the site of one excisional skin wound and six doses Placebo over the same period at the site of a second excisional skin wound. Each subject served as their own simultaneous control.
Period: Overall Study
Arm/Group | Remlarsen-Treated Excisional Skin Wound and Placebo-Treated Excisional Skin Wound
Started | 14
Completed | 12
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Remlarsen-Treated Excisional Skin Wound and Placebo-Treated Excisional Skin Wound
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Number of pre-existing keloids at screening [Mean (Standard Deviation); unit: millimeters] | 10.7 (5.44)
Height of largest pre-existing keloid [Mean (Standard Deviation); unit: millimeters] | 2.96 (3.96)
Width of largest pre-existing keloid [Mean (Standard Deviation); unit: millimeters] | 26.0 (35.0)
Length of largest pre-existing keloid [Mean (Standard Deviation); unit: millimeters] | 89.9 (83.6)
Volume of largest pre-existing keloid [Mean (Standard Deviation); unit: millimeters cubed] | 10,366 (22,607)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Confirmed Keloid Formation at Treated vs. Untreated Lesions at 24 Weeks
Description: The percentage of subjects with confirmed keloid formation at treated versus untreated lesions at 24 weeks (± 7 days) after first dose, analyzed using the modified Vancouver Scar Scale which reports a cumulative score based on subscores for vascularity, pliability and height.
Time Frame: 24 weeks (± 7 days) from first dose
Population: All subjects for whom an assessment of keloid formation using the modified Vancouver Scar Scale was performed at 24 weeks (± 7 days). Subjects who did not have keloid assessments within this time window were not included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Remlarsen-Treated Excisional Skin Wound; Placebo-Treated Excisional Skin Wound: Six doses remlarsen (5.3 mg) over a period of 2 weeks at the site of one excisional skin wound and six doses Placebo over the same period at the site of a second excisional skin wound. Each subject served as their own simultaneous control.
Arm/Group | Remlarsen-Treated Excisional Skin Wound | Placebo-Treated Excisional Skin Wound
Number analyzed (Participants) | 14 | 14
percentage of participants | 92.9 [66.13 to 99.82] | 85.7 [57.19 to 98.22]

2. Other Pre Specified Outcome: Percentage of Subjects With Improvement, Defined as no Confirmed Keloid Formation in the Treated Lesion vs. Confirmed Keloid Formation in the Untreated Lesion.
Description: Percentage of subjects with improvement at 24 weeks (± 7 days), defined as no confirmed keloid formation in the treated lesion vs. confirmed keloid formation in the untreated lesion, based on assessment using the modified Vancouver Scar Scale which reports a cumulative score based on subscores for vascularity, pliability and height.
Time Frame: 24 weeks (± 7 days) from first dose
Population: Subjects for whom an analysis of improvement, defined as no confirmed keloid formation in the treated lesion vs. confirmed keloid formation in the untreated lesion based on assessment using the modified Vancouver Scar Scale, was performed at 24 weeks (± 7 days). Subjects who did not have an analysis of improvement, as defined, were not included in this outcome measure.
Arm/Group | Remlarsen-Treated Excisional Skin Wound and Placebo-Treated Excisional Skin Wound
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Percentage of Subjects With Confirmed Keloid Formation at Treated vs. Untreated Lesions at 52 Weeks
Description: The percentage of subjects with confirmed keloid formation at treated versus untreated lesions at 52 weeks (± 7 days) after first dose, analyzed using the modified Vancouver Scar Scale which reports a cumulative score based on subscores for vascularity, pliability and height.
Time Frame: 52 weeks (± 7 days) from first dose
Population: All subjects for whom an assessment of keloid formation using the modified Vancouver Scar Scale was performed at 52 weeks (± 7 days). Subjects who did not have keloid assessments within this time window were not included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Remlarsen-Treated Excisional Skin Wound: Six doses remlarsen (5.3 mg) over a period of 2 weeks at the site of one excisional skin wound and six doses Placebo over the same period at the site of a second excisional skin wound. Each subject served as their own simultaneous control.
  Remlarsen: Intradermal injection at site of one excisional wound
- Placebo-Treated Excisional Skin Wound: Six doses remlarsen (5.3 mg) over a period of 2 weeks at the site of one excisional skin wound and six doses Placebo over the same period at the site of a second excisional skin wound. Each subject served as their own simultaneous control.
  Placebo: Intradermal injection at site of second excisional wound
Arm/Group | Remlarsen-Treated Excisional Skin Wound | Placebo-Treated Excisional Skin Wound
Number analyzed (Participants) | 6 | 6
percentage of participants | 100 [54.07 to 100.0] | 66.7 [22.28 to 95.67]

4. Other Pre Specified Outcome: Time to Keloid Formation
Description: Time to first confirmed keloid formation
Time Frame: First dose to 365 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Remlarsen-Treated Excisional Skin Wound | Placebo-Treated Excisional Skin Wound
Number analyzed (Participants) | 14 | 14
days | 58 [29 to 85] | 55 [22 to 71]

5. Other Pre Specified Outcome: Volume of Keloid at 24 Weeks
Time Frame: 24 weeks from first dose
Measure: Mean (Standard Deviation); unit: millimeters cubed
Arm/Group | Remlarsen-Treated Excisional Skin Wound | Placebo-Treated Excisional Skin Wound
Number analyzed (Participants) | 7 | 7
millimeters cubed | 65 (58) | 79 (55)

6. Other Pre Specified Outcome: Volume of Keloid at 52 Weeks
Time Frame: 52 weeks from first dose
Measure: Mean (Standard Deviation); unit: millimeters cubed
Arm/Group | Remlarsen-Treated Excisional Skin Wound | Placebo-Treated Excisional Skin Wound
Number analyzed (Participants) | 4 | 4
millimeters cubed | 194 (142) | 156 (176)

7. Other Pre Specified Outcome: Area Under the Plasma Concentration vs. Time Curve (AUC) of Remlarsen - Single Dose
Description: Area under the curve (AUClast) for remlarsen + active metabolites (total active drug) after a single dose
Time Frame: First dose to 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Remlarsen-Treated Excisional Skin Wound and Placebo-Treated Excisional Skin Wound
Number analyzed (Participants) | 14
ng*hr/mL | 461 (359)

8. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of Remlarsen - Single Dose
Description: Peak plasma concentration (Cmax) of remlarsen + active metabolites (total active drug) after first dose
Time Frame: First dose to 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Remlarsen-Treated Excisional Skin Wound and Placebo-Treated Excisional Skin Wound
Number analyzed (Participants) | 14
ng/mL | 29.3 (20.6)

9. Other Pre Specified Outcome: Area Under the Plasma Concentration vs. Time Curve (AUC) of Remlarsen - Multi-dose
Description: Area under the curve (AUClast) for remlarsen + active metabolites (total active drug) after multiple doses
Time Frame: First dose to up to 13 days post-dose
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Remlarsen-Treated Excisional Skin Wound and Placebo-Treated Excisional Skin Wound
Number analyzed (Participants) | 12
ng*hr/mL | 1200 (383)

10. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of Remlarsen - Multi-dose
Description: Peak plasma concentration (Cmax) of remlarsen + active metabolites (total active drug) after multiple doses
Time Frame: Dosing on Day 10 or Day 12 through 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Remlarsen-Treated Excisional Skin Wound and Placebo-Treated Excisional Skin Wound
Number analyzed (Participants) | 12
ng/mL | 75.5 (23.7)

ADVERSE EVENTS:
Time Frame: All adverse events from clinical trial initiation until 30 days post-dose regardless of relationship, and Related events until the end of the protocol-specified observation period.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Treatment-emergent Adverse Events, Excluding Wound or Injection-site Related Events: All subjects; all treatment-emergent adverse events, excluding wound or injection site-related events
- Wound or Injection Site-related Treatment-emergent Adverse Events: All subjects; wound or injection site-related treatment-emergent adverse events
Arm/Group | Treatment-emergent Adverse Events, Excluding Wound or Injection-site Related Events | Wound or Injection Site-related Treatment-emergent Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 12/14 | 6/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment-emergent Adverse Events, Excluding Wound or Injection-site Related Events (N=14) | Wound or Injection Site-related Treatment-emergent Adverse Events (N=14)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 5 (6)
Injection site oedema (General disorders) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Incision site pruritus (Injury, poisoning and procedural complications) | 0 (0) | 5 (6)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 4 (11) | 0 (0)
Monocyte count increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Groin infection (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators in this study may present or publish study results in scientific journals or other scholarly media without prior written approval after the following conditions have been met:

* Results of study have been publicly disclosed by or with the consent of the sponsor
* Investigator has complied with the Clinical Trial Agreement and requests from the sponsor to delete confidential information (other than study results)
* Study has been completed at all study sites for at least 2 years

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT03601052/Prot_SAP_000.pdf